CLINICAL TRIAL: NCT06833827
Title: 'Thrombectomy in High-Risk Pulmonary Embolism - Device Versus Thrombolysis Netherlands': TORPEDO-NL
Acronym: TORPEDO-NL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Zorginstituut Nederland: The Health Care Insurance Board (Unknown)
Responsible Party: Principal Investigator, Erik Klok, Clinical Professsor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL87503.058.24
Record Dates: First submitted 2025-01-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism Acute
Keywords: Acute Pulmonary Embolism; Full dose systemic thrombolysis; Catheter-directed thrombectomy
MeSH Terms: interventions — Thrombectomy; Thrombolytic Therapy; Fibrinolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Catheter-directed thrombectomy (CDT) (Experimental): Patients in the intervention group will receive Catheter-directed thrombectomy (CDT).
  Interventions: Device: Catheter-directed thrombectomy (CDT)
- Systemic Thrombolysis (Active Comparator): Patients in the control group will receive full-dose systemic thrombolysis.
  Interventions: Drug: thrombolysis therapy

INTERVENTIONS:
Device: Catheter-directed thrombectomy (CDT) — The intervention consists of immediate thrombectomy (thrombectomy with any approved device) without systemic/locally administered thrombolysis. Thrombectomy is performed via jugular or femoral venous access according to the instructions for use for the particular device. The catheter is advanced over a preplaced guidewire across the right heart into the pulmonary arteries to the location of proximal thrombus. Procedural therapeutic anticoagulation with heparin is administered. After removal of the dilator, the thrombus is extracted by controlled volume aspiration through an aspiration catheter using a syringe or dedicated aspiration system, with multiple aspirations performed as needed. Procedural objectives will be clearly stated prior to the intervention and patient's clinical and hemodynamic status and residual thrombus will guide the investigators to determine when to terminate the procedure. Treatment success is defined as clear evidence of right ventricular recompensation.
  Other Names: CDT; Thrombectomy; catheter-directed mechanical thrombectomy; mechanical thrombectomy; Catheter-based thrombectomy
  Arms: Catheter-directed thrombectomy (CDT)
Drug: thrombolysis therapy — Standard reperfusion treatment for high-risk PE patients is thrombolytic therapy, typically consisting of Alteplase, Urokinase, or Tenecteplase, with the idea of accelerated fragmentation of the thrombus by lytic medication given systemically.
  Other Names: systemic thrombolysis; full-dose systemic thrombolysis; thrombolysis; thrombolytic therapy
  Arms: Systemic Thrombolysis

SUMMARY:
TORPEDO-NL will be an investigator-initiated, academically sponsored, multicentre, open-label, randomized controlled trial (RCT).

Patients with high-risk pulmonary embolism (PE) require immediate reperfusion therapy on top of anticoagulation. The standard reperfusion treatment in these patients is full-dose systemic thrombolysis. This carries a significant risk of major bleeding (10-25%) and intracranial haemorrhage (ICH, 3%). Catheter-directed thrombectomy (CDT) is a promising alternative to systemic thrombolysis with a more direct effect on reducing pulmonary artery clot burden and very likely a better safety profile. Randomized trials evaluating the safety and efficacy of CDT in high-risk patients are currently unavailable. The investigators hypothesize that in high-risk PE patients, CDT is superior to the current standard of systemic thrombolysis in terms of mortality and adverse events, i.e., is associated with a lower composite incidence of all-cause mortality, treatment failure, major bleeding and all-cause stroke. The investigators also hypothesize that CDT will lead to a shorter length of stay (LOS) at the intensive care unit (ICU) and in-hospital, faster recovery, and better long-term quality of life (QoL).

Objective: To determine whether CDT in high-risk PE relative to systemic thrombolysis is:

* more effective and safer in terms of a reduction of the composite endpoint on all-cause mortality and adverse events defined as treatment failure, major bleeding and all-cause stroke at day 30 (primary outcome)
* leads to a better Desirability of Outcome Ranking (DOOR) at day 7
* associated with a lower level of oxygen supplementation at 48 hours
* associated with shorter length of stay (LOS) at the intensive care unit (ICU) and in the hospital
* associated with better functional recovery as well as better patient-reported outcomes such as QoL at one year
* cost-effective after a time horizon of one year

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with confirmed acute PE, i.e. contrast filling defect in a lobar or more proximal pulmonary artery on computed tomography pulmonary angiography (CTPA), and/or obstructive shock with echocardiographic confirmed dilatation of the right ventricle and a congested vena cava inferior, both with/without echocardiographic signs of clot in transit or deep vein thrombosis of the leg.
2. High risk for mortality, i.e.

   1. post cardiac arrest (after temporary need for cardiopulmonary resuscitation), OR
   2. obstructive shock (systolic blood pressure <90 mmHg and signs of end-organ hypoperfusion (e.g. elevated lactate levels >2 mmol/l) or the need for vasopressors (adrenalin or noradrenalin) to maintain an adequate blood pressure), OR
   3. persistent hypotension (systolic blood pressure <90 mmHg or systolic blood pressure drop ≥40 mmHg for at least 15 minutes) not caused by new onset arrhythmia, hypovolemia, or sepsis, OR
   4. abnormal RV function on transthoracic echocardiography or CTPA AND elevated cardiac troponin levels AND respiratory failure defined as hypoxemia (SaO2 <90%) refractory to O2 supplementation by nasal cannula or Venturi mask, requiring full face mask O2 supplementation (100% FiO2), high-flow nasal O2, or (non-)invasive mechanical ventilation.
3. CDT available and technically feasible so as to allow for a randomization-to-needle time of 60 minutes or less.

Exclusion Criteria:

1. "Catastrophic PE", i.e. ongoing cardiac arrest and/or need for extracorporeal cardiopulmonary resuscitation (ECPR) and/or immediate indication for venoarterial extracorporeal membrane oxygenation (VA-ECMO) as judged by the responsible physician(s)
2. Glascow Coma Scale <8 following resuscitation for cardiac arrest
3. Alternative diagnosis than acute PE contributing largely to the acute hemodynamic and/or respiratory failure, e.g. sepsis, COPD GOLD 3 or 4, or known heart failure with NYHA Functional Classification of 4, as judged by the treating physician.
4. A known "do not admit to the ICU" or "do not resuscitate" directive
5. An absolute contraindication to systemic thrombolysis, i.e.

   * History of hemorrhagic stroke
   * Ischemic stroke in past 6 months
   * Central nervous system neoplasm
   * Major trauma, major surgery or major head injury in past 3 weeks (note: mild external laceration of the head after, e.g. syncope, does not count as major head injury, especially when a CT scan of the head shows no hematoma)
   * Active bleeding, life-threatening or into a critically organ/area; OR known severe bleeding diathesis with previous bleeding fulfilling these criteria
6. Reperfusion therapy (systemic thrombolysis, surgical thrombectomy or CDT/other catheter directed therapy), or placement of a non-retrieved inferior vena cava filter for acute pulmonary embolism in the past 3 months
7. Thrombus in transit through a patent foramen ovale.
8. Known chronic thromboembolic pulmonary hypertension (CTEPH), or strong suspicion of CTEPH based on pre-existing clinical findings and combinations of signs of PE chronicity on echocardiography and/or CTPA.
9. Known hypersensitivity to systemic thrombolysis, heparin, or to any of the excipients
10. If, in the Investigator's opinion, or after consultation with the local PERT-team or EC-members, the patient is not appropriate for thrombectomy
11. Chronic use of full-dose oral or parenteral anticoagulation before presentation.
12. Pregnancy
13. Current participation in another study that would interfere with participation in this study
14. Previous enrolment in this study
15. Refusal of deferred consent by the next of kin or by the patient himself to use the data. Deferred consent will not be asked to relatives of patients who die in scene, but are included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The composite incidence of the binary endpoints of all-cause mortality, treatment failure, major bleeding and all-cause stroke at day 30. | Day 30
  This outcome will be assessed using patient records or information provided by the treating physician. A detailed description of treatment failure is provided in outcome 3 of the secondary outcomes. Major bleeding is defined as Bleeding Academic Research Consortium (BARC)3b and BARC3c bleeding (=intracranial haemorrhage). Ischemic stroke is defined as any stroke (National Institutes of Health Stroke Scale ≥1).
  Unit of measure: incidence (number and percentage).

SECONDARY OUTCOMES:
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a better survival. | Day 7 and day 30
  This will be assessed using patient records or information provided by the treating physician. Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower incidence of treatment failure. | Day 7 and day 30
  Treatment failure in the first six hours after randomization is defined as life-threatening hemodynamic or respiratory deterioration. This deterioration is the clinical scenario if, after randomization, the patient develops overt cardiorespiratory instability over at least 15 minutes necessitating CPR, escalation of respiratory support, or ECMO. After these first six hours, treatment failure will also be defined by increasing dosages of cardiorespiratory support (e.g. oxygen, catecholamines), and lack of improvement. Lack of improvement is defined by the presence of at least one of the following criteria: i) an equal or rising SCAI SHOCK stage, ii) an equal or rising Fraction of Inspired Oxygen (FiO2) level to maintain adequate oxygen saturation (i.e. ≥ 92%), or iii) an equal or decreasing P/F ratio.
  Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower incidence of all-cause mortality. | Day 7, day 30 and day 90
  This will be assessed using patient records or information provided by the treating physician.
  Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower incidence of all-cause stroke. | Day 7 and day 30
  Ischemic stroke is defined as any stroke (National Institutes of Health Stroke Scale ≥1).This will be assessed using patient records or information provided by the treating physician. Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower composite incidence of the binary endpoints of the primary outcome at day 7. | Day 7
  This will be assessed using patient records or information provided by the treating physician. A detailed description of treatment failure is provided in outcome 3 of the secondary outcomes. Major bleeding is defined as Bleeding Academic Research Consortium (BARC)3b and BARC3c bleeding (=intracranial haemorrhage). Ischemic stroke is defined as any stroke (National Institutes of Health Stroke Scale ≥1). Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a better Desirability of Outcome Ranking (DOOR). | Day 7
  The DOOR concept evaluates treatment benefits and harms using efficacy, safety, and functional outcomes. Patients are classified into an ordinal global outcome based on overall desirability. The probability of a more favorable result with one treatment is assessed by comparing pairwise results, ranked by the number of days requiring organ support. Organ support includes respiratory (high-flow nasal cannula or (non-)invasive mechanical ventilation) or cardiovascular (vasopressors or inotropes). DOOR outcomes, ranked from most to least desirable: 1. Survival with no severe functional limitations, no treatment failure, and no adverse events; 2. Survival with severe functional limitations, no adverse events or treatment failure; 3. Survival with BARC3b bleeding; 4. Survival with BARC3c bleeding or stroke; 5. Survival with treatment failure; 6. Death. Functional limitations are defined by the PVFS scale (grade 4 = severe limitations).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower incidence of BARC3b and BARC3c bleeding. | Day 7 and day 30
  Major bleeding is defined as Bleeding Academic Research Consortium (BARC)3b and BARC3c bleeding (=intracranial haemorrhage). This will be assessed using patient records or information provided by the treating physician. Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower incidence of ISTH major and non-major clinically relevant bleeding. | Day 7 and day 30
  This will be assessed using patient records or information provided by the treating physician. Unit of measure: incidence (number and percentage).
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with a lower level of oxygen supplementation. | 48 hours
  This will be assessed using patient records or information provided by the treating physician.
  Unit of measure: LO2/min
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with shorter length of stay (days) at the ICU (Intensive Care Unit) and in hospital. | Up to 1 year
  This will be assessed using patient records or information provided by the treating physician.
  Unit of measure: time in days.
To evaluate, after randomization, whether CDT in high-risk PE patients relative to systemic thrombolysis is associated with better patient-relevant outcomes such as Quality of life (QoL), functional recovery and symptom burden. | Day 7 and after 3, 6, 9 and 12 months
  This will be assessed using a selection of the questionnaires mentioned in the ICHOM Set of Patient-Centered Outcome Measures for Venous Thromboembolism. The exact questionnaires used can be found in Table 2 of the study protocol.
Cost-effectiveness analysis after a time horizon of one year and budget impact analysis | 1 Year
  This will be assessed using questionnaires, the exact questionnaires used can be found in Table 2 of the study protocol. A more detailed description of how cost-effectiveness and budget impact will be assessed is provided in section 10.2 of the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: F. A. Klok, Prof. MD. PhD., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Arora S, Vallabhajosyula S, Aggarwal V, Basir MB, Kelly B, Atreya AR. Novel Risk Stratification and Hemodynamic Profiling in Acute Pulmonary Embolism: A Proposed Classification Inspired by Society for Cardiovascular Angiography and Intervention Shock Staging. Interv Cardiol Clin. 2023 Jul;12(3S):e1-e20. doi: 10.1016/j.iccl.2024.04.002. Epub 2024 May 25. PMID 38964819
- [Background] Kapur NK, Kanwar M, Sinha SS, Thayer KL, Garan AR, Hernandez-Montfort J, Zhang Y, Li B, Baca P, Dieng F, Harwani NM, Abraham J, Hickey G, Nathan S, Wencker D, Hall S, Schwartzman A, Khalife W, Li S, Mahr C, Kim JH, Vorovich E, Whitehead EH, Blumer V, Burkhoff D. Criteria for Defining Stages of Cardiogenic Shock Severity. J Am Coll Cardiol. 2022 Jul 19;80(3):185-198. doi: 10.1016/j.jacc.2022.04.049. PMID 35835491
- [Background] Gwozdz AM, de Jong CMM, Fialho LS, Likitabhorn T, Sossi F, Jaber PB, Hojen AA, Arcelus JI, Auger WR, Ay C, Barco S, Gazzana MB, Bayley J, Bertoletti L, Cate-Hoek AT, Cohen AT, Connors JM, Galanaud JP, Labropoulos N, Langlois N, Meissner MH, Noble S, Nossent EJ, de Leon Lovaton PP, Robert-Ebadi H, Rosovsky RP, Smolenaars N, Toshner M, Tromeur C, Wang KL, Westerlund E, de Wit K, Black SA, Klok FA. Development of an international standard set of outcome measures for patients with venous thromboembolism: an International Consortium for Health Outcomes Measurement consensus recommendation. Lancet Haematol. 2022 Sep;9(9):e698-e706. doi: 10.1016/S2352-3026(22)00215-0. PMID 36055334
- [Background] Evans SR, Rubin D, Follmann D, Pennello G, Huskins WC, Powers JH, Schoenfeld D, Chuang-Stein C, Cosgrove SE, Fowler VG Jr, Lautenbach E, Chambers HF. Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR). Clin Infect Dis. 2015 Sep 1;61(5):800-6. doi: 10.1093/cid/civ495. Epub 2015 Jun 25. PMID 26113652
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Ende-Verhaar YM, Meijboom LJ, Kroft LJM, Beenen LFM, Boon GJAM, Middeldorp S, Nossent EJ, Symersky P, Huisman MV, Bogaard HJ, Vonk Noordegraaf A, Klok FA. Usefulness of standard computed tomography pulmonary angiography performed for acute pulmonary embolism for identification of chronic thromboembolic pulmonary hypertension: results of the InShape III study. J Heart Lung Transplant. 2019 Jul;38(7):731-738. doi: 10.1016/j.healun.2019.03.003. Epub 2019 Mar 15. PMID 30962147
- [Background] Kabrhel C, Okechukwu I, Hariharan P, Takayesu JK, MacMahon P, Haddad F, Chang Y. Factors associated with clinical deterioration shortly after PE. Thorax. 2014 Sep;69(9):835-42. doi: 10.1136/thoraxjnl-2013-204762. Epub 2014 May 20. PMID 24846902
- [Background] Pancani R, Villari L, Aquilini F, Palla A, Carrozzi L, Celi A. Prognostic role of respiratory failure in acute pulmonary embolism: a prospective multicenter study. Thromb Res. 2022 Sep;217:33-35. doi: 10.1016/j.thromres.2022.07.002. Epub 2022 Jul 9. No abstract available. PMID 35849919
- [Background] Ergan B, Ergun R, Caliskan T, Aydin K, Tokur ME, Savran Y, Koca U, Comert B, Gokmen N. Mortality Related Risk Factors in High-Risk Pulmonary Embolism in the ICU. Can Respir J. 2016;2016:2432808. doi: 10.1155/2016/2432808. Epub 2016 Nov 29. PMID 28025592
- [Background] Koslow M, Epstein Shochet G, Fenadka F, Neuman Y, Osadchy A, Shitrit D. Systemic Thrombolysis Therapy is Associated With Improved Outcomes Among Patients With Acute Pulmonary Embolism and Respiratory Failure. Am J Med Sci. 2020 Aug;360(2):129-136. doi: 10.1016/j.amjms.2020.04.028. Epub 2020 Apr 28. PMID 32466857
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Background] Huisman MV, Barco S, Cannegieter SC, Le Gal G, Konstantinides SV, Reitsma PH, Rodger M, Vonk Noordegraaf A, Klok FA. Pulmonary embolism. Nat Rev Dis Primers. 2018 May 17;4:18028. doi: 10.1038/nrdp.2018.28. PMID 29770793
- [Derived] Stenger WJE, den Uil CA, Rietdijk WJR, Al Amri I, Montero-Cabezas JM, Elzo Kraemer CV, van Mens TE, Meuwese CL, van Mieghem NMDA, Lauw MN, van den Toorn LM, Levolger S, van de Luijtgaarden KM, Sprenger RA, van Dongen JM, Imani F, Meuwissen M, Kant KM, Aarts RAHM, Winckers K, Brans RJB, Kuiper GJAJM, Schnabel R, Ende-Verhaar YM, Urlings TAJ, Ruys TA, Slot S, Scheffer HJ, Adriaansens SOJH, Boomsma MF, Nijholt IM, Walen S, Leentjens J, Jenniskens S, van Geuns RJ, Griffioen A, Nijkeuter M, Ruigrok D, Vos JA, Kies DA, Tuinman PR, Lely RJ, van der Meijs BB, Hovens MMC, Konstantinides SV, Mol MS, Kraaijeveld AO, Klok FA; Contributing authors. Thrombectomy in high-risk pulmonary embolism - device versus thrombolysis: rationale and design of the TORPEDO-NL investigator-initiated, academically-sponsored, multicenter, open-label randomized controlled trial. Thromb Res. 2025 Nov;255:109420. doi: 10.1016/j.thromres.2025.109420. Epub 2025 Aug 7. PMID 41027123

DOCUMENTS (1):
  • Study Protocol (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT06833827/Prot_000.pdf